CLINICAL TRIAL: NCT06733051
Title: A Single-arm, Open-label, Phase II Study of Golidocitinib and Benmelstobart Combination Treatment in Patients with Relapsed or Refractory Extranodal Natural Killer/T Cell Lymphoma (ENKTL) (JACKPOT50)
Brief Title: Phase II Study of Golidocitinib and Benmelstobart in Patients with R/R ENKTL (JACKPOT50)
Acronym: JACKPOT50
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, MD. PhD., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-736-01
Record Dates: First submitted 2024-12-08; First posted 2024-12-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Natural Killer T-cell Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Golidocitinib and Benmelstobart Combination (Experimental): Patients will receive golidocitinib in combination with benmelstobart every 3 weeks for up to 24 months, until disease progression, unaccpetable toxicities or other reasons lead to discontinuation.
  Interventions: Drug: Golidocitinib; Drug: Benmelstobart

INTERVENTIONS:
Drug: Golidocitinib — 150 mg, administered once daily from Day 1 to Day 21 (D1-D21)
Drug: Benmelstobart — 1200 mg, administered on Day 1 (D1) of every cycle

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial to evaluate the efficacy and safety of golidocitinib and benmelstobart combination treatment in patients with relapsed or refractory extranodal natural killer/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent.
2. Pathologically confirmed extranodal natural killer/T cell lymphoma (ENKTL).
3. Age ≥18, no gender limitation.
4. Treatment failure to at least one line of asparaginase-based therapy.
5. Eastern Cooperative Oncology Group performance status of 0-2
6. Expected survival ≥ 3 months.
7. At least one measurable lesion that meets Lugano 2014 criteria.
8. Sufficient organ function.

Exclusion Criteria:

1. Invasive NK-cell leukemia or NKTCL that has progressed to leukemia.
2. Accompanied by hemophagocytic lymphohistiocytosis.
3. NKTCL with central nervous system invasion.
4. Previously treated with JAK inhibitors.
5. The patients have contraindications to any drug in the combined treatment.
6. Patients with the infection of human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome.
7. Inability to swallow tablets, presence of malabsorption syndrome, or any other gastrointestinal disease or dysfunction that may affect the absorption of the study drug.
8. Pregnant and lactating women and subjects of childbearing age who do not want to use contraception.
9. Mentally ill persons or persons unable to obtain informed consent. The investigators think that the patient is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 2 years
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) as the best response.

SECONDARY OUTCOMES:
Complete Response(CR) | 2 years
  Defined as the proportion of patients who achieve complete remission as the best response
Duration of Response(DOR) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival(PFS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Incidence and severity of adverse events (AE) , Serious adverse event (SAE) and immune-related adverse event (irAE) | Through study completion, up tp 2 years.
  To identify the incidence of AE, SAE, and irAE.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided